CLINICAL TRIAL: NCT03980522
Title: An Open-Label Pilot Study of KPL-914 in Recurrent Pericarditis
Brief Title: A Pilot Study of KPL-914 in Recurrent Pericarditis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals (UK), Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kiniksa Pharmaceuticals International, plc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPL-914-C001
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Recurrent Pericarditis
MeSH Terms: conditions — Pericarditis | interventions — rilonacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- KPL-914: Part 1 Participants (Experimental): Part 1 enrolls symptomatic participants with recurrent idiopathic pericarditis (RIP) with an elevated marker of systemic inflammation (C-reactive protein [CRP] > 1mg/dL).
  Interventions: Drug: KPL-914
- KPL-914: Part 2 Participants (Experimental): Part 2 enrolls symptomatic participants with RIP with CRP ≤1 mg/dL which, in the opinion of the Investigator, can be attributed to concomitant medications (e.g., corticosteroids) and with pericardial inflammation present on cardiac magnetic resonance imaging (MRI) confirmed by the imaging core lab.
  Interventions: Drug: KPL-914
- KPL-914: Part 3 Participants (Experimental): Part 3 enrolls participants with corticosteroid-dependent RIP not experiencing symptoms which would meet the diagnostic criteria for a flare of pericarditis.
  Interventions: Drug: KPL-914
- KPL-914: Part 4 Participants (Experimental): Part 4 enrolls symptomatic participants with recurrent post pericardiotomy syndrome (PPS) with an elevated marker of systemic inflammation (CRP > 1mg/dL).
  Interventions: Drug: KPL-914
- KPL-914: Part 5 Participants (Experimental): Part 5 enrolls participants with corticosteroid-dependent recurrent PPS not experiencing symptoms which would meet the diagnostic criteria for a flare of pericarditis.
  Interventions: Drug: KPL-914

INTERVENTIONS:
Drug: KPL-914 — KPL-914 (rilonacept) will be provided in its commercially available formulation as a lyophilized powder to be reconstituted for SC administration.
  Adult participants (≥ 18 years of age) KPL-914 will be administered as an initial loading dose of 320 mg SC, delivered as 2 subcutaneous injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Pediatric participants (6 to <18 years of age) KPL-914 will be administered with an initial loading dose of 4.4 mg/kg, up to a maximum of 320 mg, delivered as 2 subcutaneous injections of 2.2 mg/kg each with a maximum single-injection volume of 2 mL.
  Participants considered to be 'treatment responders' will be offered participation in an optional 18-week extension period (EP) in which KPL-914 can be continued for a total duration of KPL-914 treatment of up to 24 weeks.
  Other Names: rilonacept

SUMMARY:
The purpose of this study is to assess the preliminary efficacy and safety of KPL-914 treatment in participants with recurrent pericarditis.

DETAILED DESCRIPTION:
This is an open-label, single-arm pilot study to explore clinical and biochemical endpoints of pericarditis symptomatology and to collect data to assess inter- and intra-subject variability on both at-baseline and on-treatment parameters. This study consists of 5 distinct Parts, and all participants will be treated with once-weekly subcutaneously (SC)-administered injections of KPL-914.There is an optional 18-week extension period.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Has given consent (or assent, if applicable) and signed an Informed Consent Form (ICF) (or informed assent form, if applicable).
* Male or female, of any ethnic origin.
* 6 to 75 years of age, inclusive.
* If used, has received non-steroidal anti-inflammatory drugs (NSAIDs), and/or colchicine and/or corticosteroids (in any combination) at stable dose levels for at least 7 days prior to study drug dosing (although stable doses for a shorter period will be acceptable if in the opinion of the Investigator, in consultation with the Sponsor, a shorter period of stability is not anticipated to alter the baseline CRP values) and is anticipated to continue these concomitant medications at these dose levels for the duration of the active Treatment Period.
* If female of child-bearing potential, must be nonpregnant and nonlactating and must agree to use an effective method of contraception, e.g., hormonal contraception or double-barrier birth control.
* Is able to adequately maintain a medication diary.
* Agrees to refrain from making any new, major life-style changes that may affect pericarditis symptoms (e.g., starting a new diet or changing exercise pattern) from the time of signature of the ICF (or informed assent form, if applicable) to the End-of-Trial Visit.

Parts 1, 2 and 4:

Subjects eligible for Parts 1, 2 and 4 have to present during a symptomatic episode of recurrent idiopathic pericarditis (RIP; Parts 1 and 2) and post pericardiotomy syndrome (PPS; Part 4) and a history of at least one pericarditis recurrence. They can be enrolled into Part 1 or 4 if the CRP value at screening is >1 mg/dL, and into Part 2 if a CRP ≤1 mg/dL (attributed to concomitant medications e.g., corticosteroids), and there is an evidence of pericardial inflammation on cardiac MRI confirmed by the imaging core lab.

Enrollment into Part 3 and 5:

Subjects eligible for Part 3 of this study have to present with corticosteroid-dependent RIP or PPS and history of at least 2 pericarditis recurrences.

Exclusion Criteria for All Participants:

* Has a diagnosis of pericarditis that was secondary to specific excluded etiologies, including tuberculous, neoplastic, or purulent etiologies, post-myocardial infarction (early or late), thoracic trauma, myocarditis, or systemic diseases including autoinflammatory diseases, autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.).
* Has a history of immunodepression, including a positive human immunodeficiency virus test result.
* Has received treatment within the 6-month period before dosing with any systemic immunosuppressants (other than, for example, corticosteroids or mycophenolate) which, in the opinion of the Investigator (in consultation with the Sponsor), may interfere with the study endpoints.
* Currently receiving other interleukin (IL)-1 or IL-6 blockers, Janus-activating kinase (JAK) or tumor necrosis factor (TNF) inhibitors.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations Study Director, Study Director — Kiniksa Pharmaceuticals (UK), Ltd.
Locations (14):
- United States (14):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Avail Clinical Research, LLC, DeLand, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Affinity Clinical Research Institute, Oak Brook, Illinois
  - Franciscan Physician Network Indiana Heart Physicians Cardiovascular Research Program, Indianapolis, Indiana
  - Research Integrity, LLC, Owensboro, Kentucky
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Ellipsis Research Group, Brooklyn, New York
  - Cleveland Clinic, Cleveland, Ohio
  - BI Research Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Result] Klein AL, Lin D, Cremer PC, Nasir S, Luis SA, Abbate A, Ertel A, LeWinter M, Beutler A, Fang F, Paolini JF. Efficacy and safety of rilonacept for recurrent pericarditis: results from a phase II clinical trial. Heart. 2020 Nov 23;107(6):488-96. doi: 10.1136/heartjnl-2020-317928. Online ahead of print. PMID 33229362
- [Derived] Lin D, Klein A, Cella D, Beutler A, Fang F, Magestro M, Cremer P, LeWinter MM, Luis SA, Abbate A, Ertel A, Litcher-Kelly L, Klooster B, Paolini JF. Health-related quality of life in patients with recurrent pericarditis: results from a phase 2 study of rilonacept. BMC Cardiovasc Disord. 2021 Apr 21;21(1):201. doi: 10.1186/s12872-021-02008-3. PMID 33882846

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 26 participants were enrolled in the study; however, only 25 unique participants were included in the analyses, as one participant was enrolled a second time.
Groups:
- KPL-914: Part 1 Participants: Symptomatic participants with recurrent idiopathic pericarditis (RIP) with an elevated marker of systemic inflammation (C-reactive protein [CRP] > 1 mg/dL) received KPL-914, administered as an initial loading dose of 320 mg subcutaneous (SC), delivered as 2 subcutaneous (SC) injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week extension period (EP) in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- KPL-914: Part 2 Participants: Symptomatic participants with RIP with CRP ≤ 1 mg/dL which, in the opinion of the Investigator, can be attributed to concomitant medications (e.g., corticosteroids) and with pericardial inflammation present on cardiac magnetic resonance imaging (MRI) confirmed by the imaging core lab received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- KPL-914: Part 3 Participants: Participants with corticosteroid-dependent RIP not experiencing symptoms which would meet the diagnostic criteria for a flare of pericarditis received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- KPL-914: Part 4 Participants: Symptomatic participants with recurrent post pericardiotomy syndrome (PPS) with an elevated marker of systemic inflammation (CRP > 1 mg/dL) received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- KPL-914: Part 5 Participants: Participants with corticosteroid-dependent recurrent PPS not experiencing symptoms which would meet the diagnostic criteria for a flare of pericarditis received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
Period: Treatment Period
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 3 Participants | KPL-914: Part 4 Participants | KPL-914: Part 5 Participants
Started | 13 | 3 | 6 | 1 | 3
Completed | 12 | 3 | 6 | 1 | 3
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 3 Participants | KPL-914: Part 4 Participants | KPL-914: Part 5 Participants
Started | 12 | 3 | 5 (1 participant did not sign the optional Extension Period consent form.) | 1 | 3
Completed | 12 | 3 | 5 | 1 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of study drug.
Groups:
- KPL-914: Part 1 Participants: Symptomatic participants with RIP with an elevated marker of systemic inflammation (CRP > 1 mg/dL) received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- KPL-914: Part 2 Participants: Symptomatic participants with RIP with CRP ≤ 1 mg/dL which, in the opinion of the Investigator, can be attributed to concomitant medications (e.g., corticosteroids) and with pericardial inflammation present on cardiac MRI confirmed by the imaging core lab received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- KPL-914: Part 4 Participants: Symptomatic participants with recurrent PPS with an elevated marker of systemic inflammation (CRP > 1 mg/dL) received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 3 Participants | KPL-914: Part 4 Participants | KPL-914: Part 5 Participants | Total
Number analyzed (Participants) | 12 | 3 | 6 | 1 | 3 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (10.23) | 42.7 (15.01) | 51.3 (7.84) | 34.0 (NA) — 1 participant in this arm | 42.0 (7.21) | 42.8 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 2 | 0 | 1 | 15
  Male | 3 | 0 | 4 | 1 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 3 | 6 | 1 | 3 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 2 | 1 | 0 | 0 | 0 | 3
  White | 10 | 2 | 6 | 1 | 3 | 22
Pain Rating Scale Score [Mean (Standard Deviation); unit: units on a scale] — Average level of pericarditis pain over previous 24 hours was assessed by participants at Baseline using 11-point pain Numerical Rating Scale (NRS), where "0" indicates "no pain" and "10" indicates pain "as bad as it could be."
  units on a scale | 4.6 (1.68) | 4.7 (3.06) | 1.2 (0.75) | 4.0 (NA) — 1 participant in this arm. | 2.0 (2.65) | 3.4 (2.27)

OUTCOME MEASURES:

1. Primary Outcome: Parts 1, 2 and 4: Pretreatment C-Reactive Protein (CRP) Levels
Time Frame: Screening Visit 1 (Day -3 to Day 0), Screening Visit 2 (Day -3 to Day 0), Day 0, Baseline (defined as the last non-missing assessment prior to the first study drug administration)
Population: Modified Intent-to-Treat (mITT) Population: all participants who received at least one dose of study drug. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 4 Participants
Number analyzed (Participants) | 12 | 3 | 1
mg/dL
  Screening Visit 1: number analyzed (Participants) | 11 | 2 | 0
  Screening Visit 1 | 5.921 (5.3423) | 0.645 (0.4313) |
  Screening Visit 2: number analyzed (Participants) | 2 | 0 | 0
  Screening Visit 2 | 4.455 (0.4455) |  |
  Day 0: number analyzed (Participants) | 9 | 1 | 1
  Day 0 | 5.156 (6.4150) | 0.090 (NA) — 1 participant in this arm at this time point | 1.140 (NA) — 1 participant in this arm at this time point
  Baseline | 4.907 (5.7686) | 0.460 (0.4424) | 1.140 (NA) — 1 participant in this arm at this time point
Statistical Analysis 1: Comparison: KPL-914: Part 1 Participants; Inter-subject variability of CRP levels for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of inter-subject variance and standard deviation (SD) from a mixed model for repeated measures with CRP level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled pre-baseline visits was used; Test type: Other; Inter-subject variance = 19.1908
Statistical Analysis 2: Comparison: KPL-914: Part 2 Participants; Inter-subject variability of CRP levels for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of inter-subject variance and SD from a mixed model for repeated measures with CRP level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled pre-baseline visits was used; Test type: Other; Inter-subject variance = 0.0018
Statistical Analysis 3: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 1, analysis 2]; Test type: Other; Inter-subject variance = 0.0000
Statistical Analysis 4: Comparison: KPL-914: Part 1 Participants; Intra-subject variability of CRP levels for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of intra-subject variance and SD from a mixed model for repeated measures with CRP level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled pre-baseline visits was used; Test type: Other; Intra-subject variance = 12.6852
Statistical Analysis 5: Comparison: KPL-914: Part 2 Participants; [analysis description as in outcome 1, analysis 4]; Test type: Other; Intra-subject variance = 0.1842
Statistical Analysis 6: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 1, analysis 4]; Test type: Other; Intra-subject variance = 1.0000

2. Primary Outcome: Parts 1, 2 and 4: On-Treatment Change From Baseline Over Time in CRP Levels
Time Frame: Baseline, Treatment Period (TP) Weeks 2, 3, 4, 5, 6, TP Interval Evaluation (between Weeks 3-4), End of TP (up to Week 6), Extension Period (EP): Months 1, 2, 3, 4, EP Interval Evaluation (between Weeks 15-20), Final Visit (up to Week 25)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 4 Participants
Number analyzed (Participants) | 12 | 3 | 1
mg/dL
  Change at TP Week 2: number analyzed (Participants) | 10 | 3 | 1
  Change at TP Week 2 | -5.202 (6.0296) | -0.277 (0.2538) | -1.040 (NA) — 1 participant in this arm at this time point
  Change at TP Week 3 | -4.658 (5.8115) | -0.310 (0.4246) | -1.110 (NA) — 1 participant in this arm at this time point
  Change at TP Interval Evaluation Visit: number analyzed (Participants) | 6 | 1 | 0
  Change at TP Interval Evaluation Visit | -6.937 (7.2968) | -0.090 (NA) — 1 participant in this arm at this time point |
  Change at TP Week 4: number analyzed (Participants) | 7 | 2 | 1
  Change at TP Week 4 | -2.213 (2.8854) | -0.445 (0.5445) | -1.110 (NA) — 1 participant in this arm at this time point
  Change at TP Week 5: number analyzed (Participants) | 11 | 3 | 1
  Change at TP Week 5 | -5.091 (5.9903) | -0.183 (0.2656) | -1.090 (NA) — 1 participant in this arm at this time point
  Change at TP Week 6: number analyzed (Participants) | 6 | 2 | 1
  Change at TP Week 6 | -3.805 (4.7420) | 0.090 (0.2121) | -1.060 (NA) — 1 participant in this arm at this time point
  Change at End of TP: number analyzed (Participants) | 11 | 1 | 1
  Change at End of TP | -3.987 (5.8107) | -0.040 (NA) — 1 participant in this arm at this time point | -0.610 (NA) — 1 participant in this arm at this time point
  Change at EP Month 1: number analyzed (Participants) | 10 | 3 | 1
  Change at EP Month 1 | -5.157 (6.3116) | -0.127 (0.3980) | -1.110 (NA) — 1 participant in this arm at this time point
  Change at EP Month 2: number analyzed (Participants) | 9 | 3 | 1
  Change at EP Month 2 | -3.482 (3.8944) | -0.230 (0.4973) | -1.080 (NA) — 1 participant in this arm at this time point
  Change at EP Month 3: number analyzed (Participants) | 6 | 3 | 1
  Change at EP Month 3 | -5.518 (7.6716) | -0.160 (0.3122) | -1.080 (NA) — 1 participant in this arm at this time point
  Change at EP Month 4: number analyzed (Participants) | 10 | 3 | 1
  Change at EP Month 4 | -5.267 (6.3316) | -0.150 (0.3995) | -1.070 (NA) — 1 participant in this arm at this time point
  Change at EP Interval Evaluation Visit: number analyzed (Participants) | 7 | 0 | 0
  Change at EP Interval Evaluation Visit | -7.336 (6.5875) |  |
  Change at EP Final Visit: number analyzed (Participants) | 11 | 3 | 1
  Change at EP Final Visit | -5.035 (6.0430) | -0.137 (0.3384) | -1.090 (NA) — 1 participant in this arm at this time point
Statistical Analysis 1: Comparison: KPL-914: Part 1 Participants; Inter-subject variability of CRP levels for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of inter-subject variance and SD from a mixed model for repeated measures with change from baseline in CRP level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled post-baseline visits was used; Test type: Other; Inter-subject variance = 34.1446
Statistical Analysis 2: Comparison: KPL-914: Part 2 Participants; [analysis description as in outcome 2, analysis 1]; Test type: Other; Inter-subject variance = 0.1326
Statistical Analysis 3: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 2, analysis 1]; Test type: Other; Inter-subject variance = 0.0000
Statistical Analysis 4: Comparison: KPL-914: Part 1 Participants; Intra-subject variability of CRP levels for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of intra-subject variance and SD from a mixed model for repeated measures with change from baseline in CRP level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled post-baseline visits was used; Test type: Other; Intra-subject variance = 0.0548
Statistical Analysis 5: Comparison: KPL-914: Part 2 Participants; [analysis description as in outcome 2, analysis 4]; Test type: Other; Intra-subject variance = 0.0134
Statistical Analysis 6: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 2, analysis 4]; Test type: Other; Intra-subject variance = 1.0000

3. Primary Outcome: Parts 1, 2 and 4: Pretreatment Pain NRS Scores
Description: The average level of pericarditis pain over previous 24 hours was assessed by participants at each visit using 11-point pain NRS (where "0" indicates "no pain" and "10" indicates pain "as bad as it could be").
Time Frame: Prescreening, Screening Visit 1 (Day -3 to Day 0), Screening Visit 2 (Day -3 to Day 0), Day 0, Baseline (defined as the last non-missing assessment prior to the first study drug administration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 4 Participants
Number analyzed (Participants) | 12 | 3 | 1
score on a scale
  Prescreening: number analyzed (Participants) | 2 | 2 | 0
  Prescreening | 3.0 (1.41) | 4.5 (3.54) |
  Screening Visit 1: number analyzed (Participants) | 12 | 2 | 1
  Screening Visit 1 | 4.3 (2.09) | 6.0 (2.83) | 4.0 (NA) — 1 participant in this arm at this time point
  Screening Visit 2: number analyzed (Participants) | 6 | 1 | 0
  Screening Visit 2 | 4.8 (2.23) | 4.0 (NA) — 1 participant in this arm at this time point |
  Day 0: number analyzed (Participants) | 4 | 1 | 0
  Day 0 | 4.5 (1.00) | 2.0 (NA) — 1 participant in this arm at this time point |
  Baseline | 4.6 (1.68) | 4.7 (3.06) | 4.0 (NA) — 1 participant in this arm at this time point
Statistical Analysis 1: Comparison: KPL-914: Part 1 Participants; Inter-subject variability of NRS Scores for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of inter-subject variance and SD from a mixed model for repeated measures with NRS level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled pre-baseline visits was used; Test type: Other; Inter-subject variance = 2.8139
Statistical Analysis 2: Comparison: KPL-914: Part 2 Participants; [analysis description as in outcome 3, analysis 1]; Test type: Other; Inter-subject variance = 6.9999
Statistical Analysis 3: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 3, analysis 1]; Test type: Other; Inter-subject variance = 0.0000
Statistical Analysis 4: Comparison: KPL-914: Part 1 Participants; Intra-subject variability of NRS Scores for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of intra-subject variance and SD from a mixed model for repeated measures with NRS level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled pre-baseline visits was used; Test type: Other; Intra-subject variance = 0.9693
Statistical Analysis 5: Comparison: KPL-914: Part 2 Participants; [analysis description as in outcome 3, analysis 4]; Test type: Other; Intra-subject variance = 0.0000
Statistical Analysis 6: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 3, analysis 4]; Test type: Other; Intra-subject variance = 1.000

4. Primary Outcome: Parts 1, 2 and 4: On-Treatment Change From Baseline Over Time in Pain NRS Scores
Description: as for outcome 3
Time Frame: Baseline, Treatment Period (TP) Day 3, Weeks 2, 3, TP Interval Evaluation (between Weeks 3-4), 4, 5, 6, End of TP (up to Week 6), Extension Period (EP): Months 1, 2, 3, 4, EP Interval Evaluation (between Weeks 15-20), Final Visit (up to Week 25)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 4 Participants
Number analyzed (Participants) | 12 | 3 | 1
score on a scale
  Change at TP Day 3: number analyzed (Participants) | 10 | 3 | 1
  Change at TP Day 3 | -1.7 (2.50) | -0.3 (0.58) | -3.0 (NA) — 1 participant in this arm at this time point
  Change at TP Week 2 | -3.3 (1.48) | -1.7 (1.15) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at TP Week 3 | -2.6 (1.88) | -1.0 (0.00) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at TP Interval Evaluation Visit: number analyzed (Participants) | 6 | 1 | 0
  Change at TP Interval Evaluation Visit | -3.8 (2.04) | -2.0 (NA) — 1 participant in this arm at this time point |
  Change at TP Week 4: number analyzed (Participants) | 7 | 2 | 1
  Change at TP Week 4 | -3.7 (1.60) | -1.0 (0.00) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at TP Week 5 | -3.1 (2.91) | -2.0 (1.00) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at TP Week 6: number analyzed (Participants) | 9 | 2 | 1
  Change at TP Week 6 | -3.9 (2.09) | -5.0 (4.24) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at End of TP: number analyzed (Participants) | 8 | 2 | 1
  Change at End of TP | -3.6 (1.85) | -3.0 (1.41) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at EP Month 1: number analyzed (Participants) | 10 | 3 | 1
  Change at EP Month 1 | -4.1 (1.52) | -2.0 (2.00) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at EP Month 2: number analyzed (Participants) | 10 | 3 | 1
  Change at EP Month 2 | -3.6 (2.12) | -3.7 (1.53) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at EP Month 3: number analyzed (Participants) | 7 | 3 | 1
  Change at EP Month 3 | -4.4 (1.40) | -3.7 (1.53) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at EP Month 4: number analyzed (Participants) | 10 | 3 | 1
  Change at EP Month 4 | -4.2 (1.40) | -4.7 (3.06) | -4.0 (NA) — 1 participant in this arm at this time point
  Change at EP Interval Evaluation Visit: number analyzed (Participants) | 6 | 0 | 0
  Change at EP Interval Evaluation Visit | -5.0 (1.79) |  |
  Change at EP Final Visit: number analyzed (Participants) | 11 | 3 | 1
  Change at EP Final Visit | -4.0 (1.48) | -4.7 (3.06) | -4.0 (NA) — 1 participant in this arm at this time point
Statistical Analysis 1: Comparison: KPL-914: Part 1 Participants; Inter-subject variability of NRS Scores for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of inter-subject variance and SD from a mixed model for repeated measures with change from baseline in NRS level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled post-baseline visits was used; Test type: Other; Inter-subject variance = 1.9968
Statistical Analysis 2: Comparison: KPL-914: Part 2 Participants; [analysis description as in outcome 4, analysis 1]; Test type: Other; Inter-subject variance = 0.9047
Statistical Analysis 3: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 4, analysis 1]; Test type: Other; Inter-subject variance = 0.0000
Statistical Analysis 4: Comparison: KPL-914: Part 1 Participants; Intra-subject variability of NRS Scores for Part 1, 2, and 4 participants was a designated primary endpoint. Estimates of intra-subject variance and SD from a mixed model for repeated measures with change from baseline in NRS level as the outcome, repeated effect of visit and random effect of subject. Variance Components covariance structure was assumed. The data from all scheduled post-baseline visits was used; Test type: Other; Intra-subject variance = 1.7598
Statistical Analysis 5: Comparison: KPL-914: Part 2 Participants; [analysis description as in outcome 4, analysis 4]; Test type: Other; Intra-subject variance = 2.8490
Statistical Analysis 6: Comparison: KPL-914: Part 4 Participants; [analysis description as in outcome 4, analysis 4]; Test type: Other; Intra-subject variance = 1.000

5. Primary Outcome: Parts 3 and 5: Change From Baseline Over Time in CRP Levels
Description: Baseline is defined as the last non-missing assessment prior to the first study drug administration.
Time Frame: Baseline, TP Weeks 2, 3, Interval Evaluation Visit (Weeks 3-4), 4, 5, 6, End of TP Visit (Week 6), EP Months 1, 2, 3, 4, EP Interval Evaluation Visit (Week 15-Week 20), Final Visit (up to EP Month 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | KPL-914: Part 3 Participants | KPL-914: Part 5 Participants
Number analyzed (Participants) | 6 | 3
mg/dL
  Baseline | 0.232 (0.0975) | 0.097 (0.0503)
  Change at TP Week 2: number analyzed (Participants) | 6 | 2
  Change at TP Week 2 | -0.152 (0.0857) | -0.070 (0.0424)
  Change at TP Week 3 | -0.150 (0.1158) | -0.053 (0.0404)
  Change at Interval Evaluation Visit: number analyzed (Participants) | 3 | 1
  Change at Interval Evaluation Visit | -0.183 (0.1002) | -0.100 (NA) — 1 participant in this arm at this time point
  Change at TP Week 4: number analyzed (Participants) | 3 | 2
  Change at TP Week 4 | -0.130 (0.0889) | -0.030 (0.0000)
  Change at TP Week 5 | -0.147 (0.0662) | -0.057 (0.0462)
  Change at TP Week 6: number analyzed (Participants) | 3 | 2
  Change at TP Week 6 | -0.087 (0.1861) | 0.540 (0.7212)
  Change at End of TP Visit | -0.140 (0.0822) | 0.003 (0.1305)
  Change at EP Month 1: number analyzed (Participants) | 5 | 2
  Change at EP Month 1 | -0.116 (0.1753) | -0.075 (0.0778)
  Change at EP Month 2: number analyzed (Participants) | 5 | 3
  Change at EP Month 2 | -0.124 (0.1717) | -0.007 (0.1206)
  Change at EP Month 3: number analyzed (Participants) | 2 | 2
  Change at EP Month 3 | -0.050 (0.0566) | 0.850 (1.2162)
  Change at EP Month 4: number analyzed (Participants) | 5 | 3
  Change at EP Month 4 | -0.130 (0.1147) | 0.030 (0.0656)
  Change at EP Interval Evaluation Visit: number analyzed (Participants) | 3 | 1
  Change at EP Interval Evaluation Visit | -0.160 (0.0854) | -0.100 (NA) — 1 participant in this arm at this time point
  Change at Final Visit: number analyzed (Participants) | 5 | 3
  Change at Final Visit | -0.098 (0.0841) | -0.033 (0.0586)

6. Primary Outcome: Parts 3 and 5: Change From Baseline Over Time in Pain NRS Scores
Description: The average level of pericarditis pain over previous 24 hours was assessed by participants at each visit using 11-point pain NRS (where "0" indicates "no pain" and "10" indicates pain "as bad as it could be"). Baseline is defined as the last non-missing assessment prior to the first study drug administration.
Time Frame: Baseline, TP Day 3, TP Weeks 2, 3, Interval Evaluation Visit (Weeks 3-4), 4, 5, 6, End of TP Visit (Week 6), EP Months 1, 2, 3, 4, EP Interval Evaluation Visit (Week 15-Week 20), Final Visit (up to EP Month 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPL-914: Part 3 Participants | KPL-914: Part 5 Participants
Number analyzed (Participants) | 6 | 3
score on a scale
  Baseline | 1.2 (0.75) | 2.0 (2.65)
  Change at TP Day 3: number analyzed (Participants) | 6 | 2
  Change at TP Day 3 | 0.0 (0.89) | 0.0 (0.00)
  Change at TP Week 2: number analyzed (Participants) | 6 | 2
  Change at TP Week 2 | 0.5 (1.64) | -0.5 (0.71)
  Change at TP Week 3: number analyzed (Participants) | 6 | 2
  Change at TP Week 3 | 0.3 (1.37) | -0.5 (0.71)
  Change at Interval Evaluation Visit (Weeks 3-4): number analyzed (Participants) | 3 | 1
  Change at Interval Evaluation Visit (Weeks 3-4) | 0.0 (1.00) | -1.0 (NA) — 1 participant in this arm at this time point.
  Change at TP Week 4: number analyzed (Participants) | 3 | 1
  Change at TP Week 4 | 0.7 (1.15) | 0.0 (NA) — 1 participant in this arm at this time point.
  Change at TP Week 5 | -0.3 (0.82) | 0.0 (0.00)
  Change at TP Week 6 | -0.7 (0.52) | -0.7 (0.58)
  Change at End of TP Visit (Week 6): number analyzed (Participants) | 3 | 2
  Change at End of TP Visit (Week 6) | 0.0 (0.00) | -2.5 (3.54)
  Change at EP Month 1: number analyzed (Participants) | 5 | 3
  Change at EP Month 1 | -1.0 (0.71) | -1.0 (1.00)
  Change at EP Month 2: number analyzed (Participants) | 5 | 3
  Change at EP Month 2 | -1.0 (0.71) | -1.0 (1.00)
  Change at EP Month 3: number analyzed (Participants) | 2 | 2
  Change at EP Month 3 | 0.0 (0.00) | -1.0 (1.41)
  Change at EP Month 4: number analyzed (Participants) | 5 | 3
  Change at EP Month 4 | -0.4 (1.52) | -1.0 (1.00)
  Change at EP Interval Evaluation Visit (Week 15-Week 20): number analyzed (Participants) | 3 | 1
  Change at EP Interval Evaluation Visit (Week 15-Week 20) | -1.3 (0.58) | -1.0 (NA) — 1 participant in this arm at this time point.
  Change at Final Visit: number analyzed (Participants) | 5 | 3
  Change at Final Visit | -0.6 (1.14) | -1.0 (1.00)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 25 weeks.
Groups:
- KPL-914: Part 1 Participants: Symptomatic participants with RIP with an elevated marker of systemic inflammation (CRP > 1 mg/dL) receivedKPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
- KPL-914: Part 4 Participants: Symptomatic participants with recurrent post pericardiotomy syndrome (PPS) with an elevated marker of systemic inflammation (CRP > 1mg/dL) received KPL-914, administered as an initial loading dose of 320 mg SC, delivered as 2 SC injections of 160 mg SC each on Day 0, then 160 mg SC dosed once weekly for 5 subsequent weeks.
  Participants considered to be 'treatment responders' were offered participation in an optional 18-week EP in which KPL-914 could be continued for a total duration of KPL-914 treatment of up to 24 weeks.
Arm/Group | KPL-914: Part 1 Participants | KPL-914: Part 2 Participants | KPL-914: Part 3 Participants | KPL-914: Part 4 Participants | KPL-914: Part 5 Participants
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3 | 0/6 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/3 | 0/6 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 6/6 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KPL-914: Part 1 Participants (N=12) | KPL-914: Part 2 Participants (N=3) | KPL-914: Part 3 Participants (N=6) | KPL-914: Part 4 Participants (N=1) | KPL-914: Part 5 Participants (N=3)
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KPL-914: Part 1 Participants (N=12) | KPL-914: Part 2 Participants (N=3) | KPL-914: Part 3 Participants (N=6) | KPL-914: Part 4 Participants (N=1) | KPL-914: Part 5 Participants (N=3)
Injection site reaction (General disorders) | 1 | 0 | 2 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site bruising (General disorders) | 1 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 1 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Application site bruise (General disorders) | 1 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site joint warmth (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Ulcer haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 2 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
High density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0 | 0
Lipids increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the first right to publish information obtained from the trial. After Sponsor publishes, PI may publish its own trial results, provided that Sponsor may embargo such publication for up to 60 days for purposes of identifying confidential information (other than trial data) that must be removed and up to an additional 90 days to prepare a patent application if there is patentable subject matter in the PI's proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT03980522/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT03980522/SAP_001.pdf